CLINICAL TRIAL: NCT01746654
Title: A Randomized Double-Blind Placebo-Controlled Study to Determine Safety of P128 Applied to Nares of Healthy Volunteers and Safety And Efficacy of Any Patient Including Chronic Kidney Disease Patients Who Are Nasal Carriers of S.Aureus.
Brief Title: Safety & Efficacy of an Antibacterial Protein Molecule Applied Topically to the Nostrils of Volunteers and Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GangaGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P128-001
Record Dates: First submitted 2012-12-05; First posted 2012-12-11 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Infectious Disease; Bacterial Infections
Keywords: S.aureus; Methicillin Resistant S.aureus (MRSA); Nasal carrier status; Prophylaxis
MeSH Terms: conditions — Communicable Diseases; Bacterial Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- P128-0.1 mg (Experimental): Three healthy adult volunteers will be enrolled to P128-0.1 mg single dose-cohort 1 (Part A) Three healthy adult volunteers will be enrolled to P128-0.1 mg multiple doses-Cohort 4 (Part B) Ten chronic kidney disease patients will be enrolled to P128-0.1 mg multiple doses (Part C) Ten patient harboring S.aureus nasally will be enrolled to P128-0.1 mg single dose (Part D)
  Interventions: Drug: P128-0.1 mg
- P128-0.3 mg (Experimental): Three healthy adult volunteers will be enrolled to P128-0.3 mg single dose-Cohort 2 (Part A) Three healthy adult volunteers will be enrolled to P128-0.3 mg multiple doses-Cohort 5 (Part B) Ten chronic kidney disease patients will be enrolled to P128-0.3 mg multiple doses (Part C) Ten patient harboring S.aureus nasally will be enrolled to P128-0.3 mg single dose (Part D)
  Interventions: Drug: P128-0.3 mg
- P128-1.0 mg (Experimental): Three healthy adult volunteers will be enrolled to P128-1.0 mg single dose-Cohort 3 (Part A) Three healthy adult volunteers will be enrolled to P128-1.0 mg multiple doses-Cohort 6 (Part B) Ten chronic kidney disease patients will be enrolled to P128 1.0 mg multiple doses (Part C) Ten patient harboring S.aureus nasally will be enrolled to P128-1.0 mg single dose (Part D)
  Interventions: Drug: P128-1.0 mg
- Placebo (Placebo Comparator): Three healthy adult volunteers will be enrolled to placebo single dose-Cohort 1-3 (Part A) Three healthy adult volunteers will be enrolled to placebo multiple doses-Cohort 4-6 (Part B) Ten chronic kidney disease patients will be enrolled to placebo multiple doses (Part C) Ten patient harboring S.aureus nasally will be enrolled to placebo single dose (Part D)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: P128-0.1 mg — P-128 at 0.1 mg divided evenly between the nares is administered once in Part A; multiple times in Part B and Part C; and once in Part D.
  Other Names: Single dose in Part A; Multiple doses in Part B; Multiple doses in Part C; Single dose in Part D
  Arms: P128-0.1 mg
Drug: P128-0.3 mg — P-128 at 0.3 mg divided evenly between the nares is administered once in Part A; multiple times in Part B and Part C; and once in Part D.
  Other Names: Single dose in Part A; Multiple doses in Part B; Multiple doses in Part C; Single dose in Part D
  Arms: P128-0.3 mg
Drug: P128-1.0 mg — P-128 at 1.0 mg divided evenly between the nares is administered once in Part A; multiple times in Part B and Part C; once in Part D.
  Other Names: Single dose in Part A; Multiple doses in Part B; Multiple doses in Part C; Single dose in Part D
  Arms: P128-1.0 mg
Drug: Placebo — Placebo was administered to both nares once in part A, multiple times in Part B and Part C, Once in part D
  Other Names: Single dose in Part A; Multiple doses in Part B; Multiple doses in Part C; Single dose in Part D
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the antibacterial protein P128 is (i) safe and well tolerated in healthy volunteers and in chronic kidney diseases patients on dialysis, (ii) is it effective in reducing the nasal carriage of pathogen (Staphylococcus aureus) in humans.

DETAILED DESCRIPTION:
Staphylococcus aureus with acquired multiple-drug resistance poses an increasing problem in both hospital and community settings. S. aureus is known to cause infections ranging in severity from skin infection to systemic bacteremia. As nasal colonization is the principal ecological niche for these bacteria and has been shown to be a significant risk factor in developing S. aureus infection, it is of importance to develop an efficient therapy that is able to clear this bacterium from human nostrils.

In-vivo studies have shown that P128 treatment is efficacious in reducing and decolonizing MRSA bacteria from rat nostrils.

Pre-clinical safety studies in animal models indicated no test drug related toxicity signs at the site of application or systemically.

The present clinical trial is conducted in four parts. Part A consists of safety and tolerability studies in 4 cohorts of 3 healthy subjects who are administered a single dose of three escalating concentrations of the drug and placebo intra-nasally. Part B consists of safety & tolerability as in part A but with multiple doses (3 doses/day for 5 days). Part C comprises of safety/tolerability as well as efficacy studies in chronic kidney disease patients stable on dialysis who are nasal carriers of S.aureus or MRSA on a treatment regimen as in Part B. Part D comprises of safety and efficacy studies in any patient who are nasal carriers of S.aureus or MRSA with single dose of 3 escalating concentrations of the drug and placebo intra-nasally.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human volunteer
* Any patient clinically stable who are nasal carrier of S. aureus or MRSA including Chronic Kidney disease patients stable on dialysis

Exclusion Criteria:

* Presence of active systemic bacterial infection of any nature not cured at least 4 weeks before enrollment.
* Systemic or intra-nasal anti-bacterial treatment during four week period before enrollment
* Pregnancy, breast feeding during the study duration
* Participation in any other intervention study during the past three months

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-12; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (Part A, Part B, Part C and Part D); Efficacy (Part C and Part D) | 30 Days (Part A and Part B), 20 Days (Part C), 7 Days (Part D)
  The number of adverse events, type of adverse events, frequency of adverse events and proportion of subjects with adverse events and the severity, seriousness and the relationship of adverse event to the treatment. For efficacy, rate of S. aureus clearance following 5 days of treatment with various doses of P128 for Part C; rate of clearance following single dose treatment with various doses of P128 for Part D.

SECONDARY OUTCOMES:
Immunogenicity (Part A, Part B and Part C) | 8 Days (Part A), 13 Days (Part B)
  Levels of antibodies to the investigational product in serum before and after administration of the drug will be compared to understand immunogenicity of the drug.
Pharmacokinetics (Part A and Part B) | 1 Day (Part A), 6 days (Part B)
  AUC0-t, AUC0-∞, Cmax, Tmax, Tlag, Kel and AUC_% will be measured; AUC means area under curve
  Part A Baseline Pre-dose: before 1st dose on Day 1. Post - dose: 5 min, 15 min, 30 min, 1hr, 2hrs and 6hrs after first dose(on day 1)
  Part B Baseline Pre-dose: before 1st dose on Day 1. Post - dose: 5 min, 15 min, 30 min, 1hr, 2hrs and 6hrs after first dose(on day 1) Pre-final dose Post - dose: 5 min, 15 min, 30 min, 1 hr, and 12 hours post last dose - after the last dose is administered.
Secondary efficacy (Part C) | 3 days
  Rate of S. aureus clearance following 3 days of treatment with various doses of P128
Re-colonization (Part C) | 14 Days
  Rate of re-colonization by S. aureus 7 and 14 days after the last day of treatment with various doses of P128

CONTACTS AND LOCATIONS:
Overall Officials: Dale A Fisher, MBBS, FRACP, Principal Investigator — National University Hospital, Singapore; Surinder Kher, MD, Study Director — Manipal Acunova Ltd, Bangalore
Locations (1):
- National University Hospital, Singapore, Singapore